CLINICAL TRIAL: NCT02757612
Title: Study Evaluating the Laser Diode Effect on Burning Mouth Syndrome
Brief Title: Study Evaluating the Laser Diode Effect Burning Mouth Syndrome
Acronym: laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Pia Lopez Jornet, MD,DDS,PhD, Universidad de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVERSIDAD DE MURCIA
Record Dates: First submitted 2016-04-27; First posted 2016-05-02 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Burning Mouth Syndrome
Keywords: laser diode, pain
MeSH Terms: conditions — Burning Mouth Syndrome; Pain | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Active Comparator): Device Laser diode parameters: spot size of 0.04 mm2, average power (output) of 40 mW and 0.4 J per irradiation point, energy density of 10 J cm2, irradiation time of 10 seconds per point
  1 session per week during 4 session
  Interventions: Radiation: laser diode
- Comparator (Sham Comparator): laser probe inactive for similar duration as for the laser diode group; only a beep sound was produced by the laser machine
  1 session per week during 4 session
  Interventions: Radiation: laser diode

INTERVENTIONS:
Radiation: laser diode — laser diode

SUMMARY:
The aim of this study was to report the effect of laser diode on the treatment of burning mouth syndrome (BMS)

Patients were randomly allocated to two different groups:

the first one (group A) underwent Laser diode whereas the second one (group B) received Laser diode inactive

DETAILED DESCRIPTION:
The inclusion criteria were as follows: (a) oral burning sensation, at least in the last 6 months; (b) no detection of oral mucosal lesions; and (c) ability to complete the present clinical trial. The exclusion criteria were as follows: (a) diagnosis of Sjögren syndrome on the basis of European criteria ; (b) previous head and neck radiotherapy; (c) diagnosed lymphoma; (d) hepatitis C infection; (c) pregnant or breast-feeding women

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of burning mouth syndrome in accordance the International Classification of Headaches: continuous symptoms of oral burning or pain on a daily or almost daily basis, during all or part of the day for more than 6 months

Exclusion Criteria:

* history of head and neck malignancy, radiation therapy to the head and neck area, poorly managed diabetes mellitus, chronic thyroid disease, or known Sjogren's disease and pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Pain | 4 weeks
  VAS (Visual Analog Scale).

SECONDARY OUTCOMES:
xerostomia | 4 weeks
  Xerostomia severity test (Xerostomia Inventory):
oral quality of life | 4 weeks
  Oral Health Impact Profile (OHIP-14)
anxiety and depression | 4 weeks
  Levels of anxiety and depression were assessed by Hospital Anxiety and Depression Scale (HADS

CONTACTS AND LOCATIONS:
Overall Officials: Lopez-Jornet Pia, MD DDS PhD, Principal Investigator — University Murcia
Locations (1):
- Pia Lopez Jornet, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loncar B, Stipetic MM, Baricevic M, Risovic D. The effect of low-level laser therapy on salivary glands in patients with xerostomia. Photomed Laser Surg. 2011 Mar;29(3):171-5. doi: 10.1089/pho.2010.2792. Epub 2010 Nov 6. PMID 21054200
- [Background] Arduino PG, Cafaro A, Garrone M, Gambino A, Cabras M, Romagnoli E, Broccoletti R. A randomized pilot study to assess the safety and the value of low-level laser therapy versus clonazepam in patients with burning mouth syndrome. Lasers Med Sci. 2016 May;31(4):811-6. doi: 10.1007/s10103-016-1897-8. Epub 2016 Feb 12. PMID 26873501
- [Background] Spanemberg JC, Lopez Lopez J, de Figueiredo MA, Cherubini K, Salum FG. Efficacy of low-level laser therapy for the treatment of burning mouth syndrome: a randomized, controlled trial. J Biomed Opt. 2015 Sep;20(9):098001. doi: 10.1117/1.JBO.20.9.098001. PMID 26359814
- [Background] Pezelj-Ribaric S, Kqiku L, Brumini G, Urek MM, Antonic R, Kuis D, Glazar I, Stadtler P. Proinflammatory cytokine levels in saliva in patients with burning mouth syndrome before and after treatment with low-level laser therapy. Lasers Med Sci. 2013 Jan;28(1):297-301. doi: 10.1007/s10103-012-1149-5. Epub 2012 Jul 8. PMID 22773117